CLINICAL TRIAL: NCT05423080
Title: Comparison of Anesthetic Induction Time and Change of Bispectral Index Between Intravenous Bolus Administration and Continuous Infusion of Remimazolam for Anesthetic Induction: a Prospective Randomized Single-blind Study
Brief Title: Anesthesia Induction With Intravenous Bolus or Continuous Infusion of Remimazolam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Hana Pharm Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Byung Gun Lim, Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022GR0114
Record Dates: First submitted 2022-06-09; First posted 2022-06-21 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Adult; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bolus group (Experimental): Participants in this group are administered remimazolam via the bolus injection method during anesthesia induction.
  Interventions: Drug: Bolus injection of remimazolam
- Infusion group (Active Comparator): Participants in this group are administered remimazolam via the continuous infusion method during anesthesia induction.
  Interventions: Drug: Infusion of remimazolam

INTERVENTIONS:
Drug: Bolus injection of remimazolam — Participants in this group are administered 0.2 mg/kg remimazolam via the bolus injection method for 20 seconds during anesthesia induction. If loss of consciousness (LOC) does not occur, the investigators will administer additional doses of 0.05 mg/kg repeatedly until LOC occurs.
  Other Names: Bolus injection of Byfavo
  Arms: Bolus group
Drug: Infusion of remimazolam — Participants in this group are administered remimazolam at a rate of 6 mg/kg/hr via the continuous infusion method during anesthesia induction. If loss of consciousness (LOC) does not occur, the investigators will escalate infusion dose to 12 mg/kg/hr until LOC occurs.
  Other Names: Continuous infusion of Byfavo
  Arms: Infusion group

SUMMARY:
Bolus injection and continuous infusion are two widely used methods for intravenous administration of drugs. Bolus injection possibly leads to a rather high drug plasma concentration temporarily, however, it can induce a rapid onset of drug effects and attain a desired clinical state fast. On the contrary, continuous infusion is able to avoid excessive drug levels in plasma, but it takes longer to achieve the proper effect.

In this study, the investigators hypothesize that the bolus injection of remimazolam can reduce anesthesia induction time when compared to the continuous infusion of remimazolam, and also maintain hemodynamic stability. (The researchers will investigate the effect of the bolus injection of remimazolam during anesthesia induction in terms of its safety and efficacy when compared with the continuous infusion.)

ELIGIBILITY:
Inclusion Criteria:

* Adults 19 years of age or older undergoing surgery under general anesthesia
* ASA I-III

Exclusion Criteria:

* Intraoperative regional blocks (e.g. spinal anesthesia, epidural anesthesia, peripheral nerve block)
* Liver resection or liver transplantation
* Cardiopulmonary bypass
* Uncontrolled HTN (SBP ≧180 mmHg, or ≧160 in patients taking antihypertensive drugs)
* Uncontrolled DM (HbA1c antihypertensive drugs ≧9.0%)
* Total bilirubin ≧3.0 mg/ml or AST or ALS ≧2.5 times the upper limit of normal
* Serum creatinine ≧2.0 mg/ml or ESRD on dialysis
* COPD in need of treatment
* Patients who are expected to have difficulty in tracheal extubation immediately after surgery for postoperative lung management
* Resistance to benzodiazepines
* Hypersensitivity to benzodiazepines, remifentanil, fentanyl citrate, rocuronium, sugammadex, flumazenil, or other anesthetic drugs
* Myasthenia gravis or myasthenic syndrome
* Myocardial infarction, transient ischemic attack, stroke, newly diagnosed coronary artery disease, percutaneous coronary intervention, or coronary artery bypass graft within 6 months
* Implantation of rate-responsive cardiac pacemaker with bioelectrical impedance sensor
* Organic brain disorder, or other neurologic diseases that cannot adequately measure EEG (BIS)
* Severe allergic diseases
* Cognitive impairment that makes it impossible to understand the instructions and informed consent of this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
MOAA/SS (sedation level) | From initiation of remimazolam to LOC (up to 5 minutes)
  The investigators will measure MOAA/SS from the start of remimazolam administration to loss of consciousness (LOC), and compare it between the two groups.

SECONDARY OUTCOMES:
Time from initiation of drug administration to bispectral index(BIS) <60 | From initiation of remimazolam to BIS <60 (up to 10 minutes)
  The investigators measure how long it takes from the start of remimazolam administration to reach BIS <60.
BIS | From initiation of remimazolam to 15 minutes after surgical incision
  The investigators will measure BIS from the start of remimazolam administration to 15 minutes after surgical incision.
Hemodynamic stability (i.e. blood pressure, heart rate) | From initiation of remimazolam to 15 minutes after surgical incision
  The investigators will evaluate hemodynamic stability from the start of remimazolam administration to 15 minutes after surgical incision

CONTACTS AND LOCATIONS:
Overall Officials: Byung Gun Lim, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea